CLINICAL TRIAL: NCT01465256
Title: Postpolypectomy Bleeding in Patients Undergoing Colonoscopy on Antiplatelet Therapy. - Multicenter, Prospective Observational Study -
Brief Title: Postpolypectomy Bleeding in Patients With Antiplatelet Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Gun, Kim. M.D., Ph.D., Assistant professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: KASIDPOLYP
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Bleeding Complication During Colon Polypectomy
Keywords: Aspirin; Colon polypectomy; Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Aspirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin holding group (No Intervention): Aspirin holding group (group 1): the patients enrolled into group 1 can stop taking aspirin during colon polypectomy. The patients are usually taking aspirin for primary prevention of vascular disease and have no risk of thromboembolism despite of they stop taking aspirin temporary
- Aspirin continuing group (Experimental): Aspirin continuing group (group 2): the patients enrolled into group 2 should take aspirin during colon polypectomy because these patients are usually take thienopyridines and aspirin, and if they would stop taking aspirin during colon polypectomy, they have a thromboembolism risk.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin hold for a certain period of time in the patients who take aspirin for the primary prevention of vascular disease,
  Arms: Aspirin continuing group

SUMMARY:
The purpose of this study is to determine if the use of aspirin prior to colonoscopy increases the risk of post polypectomy bleeding. The primary end point is comparison of bleeding rates after polypectomy of a continuous aspirin group and temporally aspirin-quit group. The secondary end point is analysis of risk factors which affect early or delayed post polypectomy bleeding.

DETAILED DESCRIPTION:
Based on very limited evidences, ASGE recommended that endoscopic procedures may be performed on patients taking aspirin. However in a survey of ASGE members regarding their endoscopic practice, 81% would consider discontinuation of aspirin before colonoscopy and 66% would not perform snare polypectomy if patients had not discontinued aspirin. Although a large prospective randomized control trial would be the ideal way to address this issue theoretically, the investigators hypothesized that there are no differences of the post polypectomy bleeding rate in patients whether continuous taking aspirin prior to polypectomy or not.

In this study, we classified the patients into two groups; the patients who can stop taking aspirin before colon polypectomy will be enrolled into group 1, and the patients who take both thienopyridines and aspirin for their underlying disease and should keep take aspirin during colon polypectomy will be enrolled into group 2. The patients of group 1 stop taking aspirin 7 days before polypectomy.

thromboembolism. Exclusions are as follow; patients taking anti-thrombotic agents, patients have low a platelet count (<80,000/mm3) and/or prolongated PT/aPTT, patients who have chronic renal disease (creatinine>3mg/dl over 6 months), patients who have GI malignancies, patients who are over ASA classification class III, over 2 score of HAS-BLED and over 1 of CHAD2 score. The expected enrolled patients number is 500 patients (250 in each group).

All cases of polypectomy are performed with identical methodology; resection after epinephrine mixture injection under blended or mixed current wave. The data includes the patients information such as sex, age, body weight, BMI and vascular disease history such as hypertension, diabetes, ischemic heart disease, cerebrovascular disease, COPD, modified HAS-BLED score and CHADS2 score. The data of polyp related factor include number of polyps, bleeding status(acute, early, delayed/minimal, moderate, sever), endoscopist (staff or fellow), bowel preparation status, polyp character (shape, location, pathology) and procedures for bleeding (clipping, APC, epinephrine injection, band ligation etc.).

All procedure will be performed with the endoscopist blinded to the patient status of whether the patient is taking aspirin continuously or not.

ELIGIBILITY:
Inclusion Criteria:

* The patients who take low dose aspirin (75~160mg) for primary prevention of vascular disease and low risk for thromboembolism.

Exclusion Criteria:

* The patients who taking anti-thrombotic agents,
* The patients who taking thienopyridines or other NSAID with aspirin,
* The patients who have low platelet count(<80,000/mm3) and prolongated PT/aPTT in laboratory test,
* The patients who have chronic renal disease (creatinine>3mg/dl over 6 months),
* The patients who have polyps over than 1 cm in size or thick pedicle over 1 cm,
* The patients who have GI malignancies,the patients who are over ASA classification class III.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
postpolypectomy bleeding rate | bleeding after polypectomy within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Soonchunhyang univerisity hospital, Seoul, Seoul, South Korea